CLINICAL TRIAL: NCT00786721
Title: Diffuse Optical Spectroscopy Measurement Technique is Helping Develop More Effective Diagnostic Tools and Therapeutic Regimes for Diabetes, Metabolic Syndrome and Other Mitochondrial Diseases Some Time in the Future
Brief Title: Mitochondria and Metabolic Syndrome in a Southern California Chinese Cohort
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Virginia Kimonis, MD, MRCP, University of California, Irvine
Other Study IDs: 20022608.
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Metabolic Syndrome; Type 2 Diabetes Mellitus
Keywords: Mitochondria and Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diffuse Optical Spectroscopy: muscle properties scanning
  Interventions: Device: Diffuse Optical Spectroscopy

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy — muscle properties scanning

SUMMARY:
There has been increasing support for our hypothesis that mitochondrial dysfunction plays an important role in the etiology of Type 2 Diabetes Mellitus and the overlapping Metabolic Syndrome.

DETAILED DESCRIPTION:
Once the mitochondrial defect(s) of these subjects has been defined, the data will be used to develop two non-invasive screening tools to detect mitochondrial defects in Diabetes Mellitus and Metabolic Syndrome patients.

The device call Diffuse Optical Spectroscopy develope at Beckman Laser Instituteis is non-invasive measurement technique, to measure the properties of the muscle tisuue and vascular activity (calf, bicep, or the brain)to evaluate the patient's metabolic status and and to assess muscle mitochondrial OXPHOS function.

ELIGIBILITY:
Inclusion Criteria:

* Chinese descent and have been clinically diagnosed with diabetes mellitus (DM) or have met the study criteria for metabolic syndrome (MS).

Exclusion Criteria:

* non chiness descent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic, community sample, residents in a Southern California Chinese Cohort
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2006-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Near Infrared Spectroscopy to assess muscle mitochondrial OXPHOS function. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Tromberg, PhD, Principal Investigator — Beckman Laser Institute University of California Irvine; Douglas c Wallace, PhD, Principal Investigator — UCI, Molecular and Mitochondrial medicine and Genetics
Locations (1):
- Beckman Laser Institute Medical clinic, Irvine, California, United States